CLINICAL TRIAL: NCT01395147
Title: An Open-label, Long-Term Extension Study to Assess the Safety and Efficacy of Lu AA21004 in Patients With Major Depressive Disorder (Extension to Lu AA21004/CCT-003 Study)
Brief Title: Long-Term Extension Study of Lu AA21004 in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuAA21004/OCT-001; JapicCTI-111530 (Registry Identifier: JapicCTI); U1111-1122-3910 (Registry Identifier: WHO)
Record Dates: First submitted 2011-07-11; First posted 2011-07-15 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lu AA21004 group (Experimental)
  Interventions: Drug: Lu AA21004

INTERVENTIONS:
Drug: Lu AA21004 — Lu AA21004 10 mg, tablets, orally, once daily for 2 weeks; reduced to 5 mg or increased to 20 mg, once daily if necessary according to the responses and symptoms of participants for up to 50 weeks.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Lu AA21004 in participants with major depressive disorder after completion of an 8-week double-blind treatment period in a preceding study (Lu AA21004/CCT-003; NCT01355081).

DETAILED DESCRIPTION:
Lu AA21004 was discovered by H. Lundbeck A/S, and is under co-development by H. Lundbeck A/S and Takeda for the treatment of major depressive disorder and general anxiety disorder.

Major depressive disorder (MDD) is a chronic, recurring disease with considerable morbidity in the general population. The estimated lifetime prevalence of major depression in the adult population is 5 to 25%, with approximately 2-fold higher prevalence in women than in men. The hallmark of the disease is a depressed mood, with additional symptoms including sleep disturbances, psychomotor agitation or retardation, sexual dysfunction, weight loss, concentration difficulties and delusional ideas. In addition to direct ill effects, MDD causes suicide or job loss and exerts indirect influence on social economy.

This long-term extension study will assess the safety and efficacy of 52-week treatment with Lu AA21004 in participants with major depressive disorder after completion of the 8-week double-blind treatment period in the preceding study (LuAA21004/CCT-003; NCT01355081; hereinafter referred to as CCT-003). This study will be conducted at the same institutions as CCT-003.

This study will include participants who completed the 8-week double-blind treatment period in CCT-003, and who meet all of the inclusion criteria, and do not meet any of the exclusion criteria of the long-term study. Visit 1 in this study will be the last visit (Visit 7) during the 8-week double-blind treatment period in CCT-003. Participants will start 2-week treatment with 10 mg/day of Lu AA21004 on the day after completion of the 8-week double-blind treatment period in CCT-003. The dose may then be decreased to 5 mg/day or increased to 20 mg/day according to the responses and symptoms of the participants. A dose increase, however, will be allowed only if the Clinical Global Impression (CGI) score meets the criteria for dose increases and the investigator or sub-investigator considers it necessary to increase the dose. The same dose should be maintained for at least 2 weeks after a dose change, except when immediate dose reduction is required for safety reasons. Neither dose increase from 5 to 20 mg nor dose reduction from 20 to 5 mg will be allowed.

The duration of administration will be 52 weeks. Participants will visit the study site every 2 weeks during the first month of treatment and every 4 weeks thereafter (Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52). Participants will be followed up 4 weeks after the last dose of the study drug, and those who prematurely discontinue the study will also be followed up 4 weeks after the last dose, whenever possible.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the double-blind treatment period of the preceding study (CCT-003)
2. Signs and dates a written, informed consent form for this study, different from that for the preceding study (CCT-003).
3. Has CGI-S score improved at least one point at completion of the 8-week double-blind treatment period compared to the Baseline Visit in the preceding study (CCT-003).
4. In the opinion of the investigator, the subject appears to benefit from long-term treatment of Lu AA21004.

Exclusion Criteria:

1. Diagnosed with the following disorder or symptom in the preceding study (CCT-003):

   * Any current psychiatric disorder other than MDD as defined in a Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR).
   * Any substance-related disorder (except nicotine and caffeine-related disorders) as defined in the DSM-IV-TR.
   * Clinically significant neurological disorder (including epilepsy).
   * Neurodegenerative disorder (Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington's disease, etc.).
   * Any DSM-IV-TR axis II disorder that might compromise this study.
2. Is at significant risk of suicide, or had a score ≥5 on Item 10 (suicidal thoughts) of the MADRS or attempted suicides during the preceding study (CCT-003)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Treatment-emergent Adverse Events | 52 Weeks.
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after the last dose of study drug, or if a serious adverse event, within 30 days after the last dose of study drug.
Number of Participants With Markedly Abnormal Laboratory Values | Up to week 52.
  The number of participants with any markedly abnormal standard safety laboratory values collected at weeks 4, 12, 24, 36, 48 and 52 relative to baseline.
Significant Change from Baseline in Body Weight | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52.
  Change from baseline in participant's weight measured throughout study.
Change from Baseline in Vital Signs | 52 Weeks.
  Vital signs will include body temperature (oral or tympanic measurement), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm).
Change from Baseline in Electrocardiograms | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52.
  Change from baseline in electrocardiograms measured throughout study.
Clinically Significant Change From Baseline in Physical Examination Findings | 52 Weeks.
  Physical examination consists of examinations of the following body systems: (1) eyes; (2) ears, nose, throat; (3) cardiovascular system; (4) respiratory system; (5) gastrointestinal system; (6) dermatologic system; (7) extremities; (8) musculoskeletal system; (9) nervous system; (10) lymph nodes; and (11) physical examinations other than body systems described in (1) to (10).

SECONDARY OUTCOMES:
Change from Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score at each time point | Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52.
  The change between MADRS score at week 8 or final visit relative to baseline. MADRS is a 10-item clinician rated scale that measures overall severity of depressive symptoms (i.e., apparent sadness, reported sadness, inner tension, etc.) rated on a 7-point Likert scale from 0 (normal) to 6 (most abnormal) with a total score range from 0 to 60. Higher scores indicate greater severity of symptoms.
Change from Baseline in the Clinical Global Impression Scale-Severity (CGI-S) score at each time point | Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52.
  The CGI-S assesses the clinician's impression of the subject's current state of mental illness and consists of one question for the investigator: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on a seven-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill). Higher scores indicate greater severity of illness.
Change from Baseline in the Clinical Global Impression - Improvement (CGI-I) score at each time point | Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52.
  The CGI-I assesses the clinician's impression of the subject's state of mental illness improvement and consists of one question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on a seven-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; 7=very much worse). Higher scores indicate greater severity of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Takeda
Locations (32):
- Japan (32):
  - Inzai-shi, Chiba
  - Noda, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Annaka-shi, Gunma
  - Fujioka-shi, Gunma
  - Takasaki-shi, Gunma
  - Hatsukaichi-shi, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Ibaraki, Ibaraki
  - Fujisawa-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Osaka, Kita-ku
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Kurashiki-shi, Okayama-ken
  - Osaka, Osaka
  - Fukaya-shi, Saitama
  - Saitama, Saitama
  - Utsunomiya, Tochigi
  - Anan-shi, Tokushima
  - Tokushisma-shi, Tokushima
  - Hachioji-shi, Tokyo
  - Katsushika-ku, Tokyo
  - Musashino-shi, Tokyo
  - Tokyo, Tokyo
  - Nanyo-shi, Yamagata

REFERENCES:
- [Derived] Inoue T, Nishimura A, Sasai K, Kitagawa T. Randomized, 8-week, double-blind, placebo-controlled trial of vortioxetine in Japanese adults with major depressive disorder, followed by a 52-week open-label extension trial. Psychiatry Clin Neurosci. 2018 Feb;72(2):103-115. doi: 10.1111/pcn.12623. Epub 2017 Dec 27. PMID 29160598